CLINICAL TRIAL: NCT02353364
Title: Prospective Randomised Control Trial of Blastocyst Euploidy Assessment and Conditioned Embryo Transfer for Infertility Patients of Advanced Maternal Age
Brief Title: Blastocyst Euploidy Assessment and Conditioned embryO traNsfer
Acronym: BEACON
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Dr Li Wang, PGS trial co-ordinator, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: PLA-001
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Infertility
Keywords: Advanced maternal age; Aneuploidy
MeSH Terms: conditions — Infertility; Aneuploidy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Transfer of 1 or 2 biopsied euploid embryo of high morphological grade based on NGS testing using CNV-Seq (PGS)
  Interventions: Other: PGS
- Group B (No Intervention): Transfer of 1 or 2 non-biopsied embryo of high morphological grade (no PGS)

INTERVENTIONS:
Other: PGS — Embryos screened by the validated NGS technology CNV-Seq
  Arms: Group A

SUMMARY:
The study is designed to evaluate the effectiveness of pre-implantation genetic screening (PGS) for infertility patients of advanced maternal age undergoing assisted reproductive treatment. Half of the patients will have their embryos tested by PGS and 1 or 2 chromosomally normal embryos with the highest morphological grading transplanted back to the uterus. The other half of the participants will not have their embryos tested and 1 or 2 untested embryos with the highest morphological grading transplanted back to the uterus.

DETAILED DESCRIPTION:
PGS is an assisted reproductive technology that screens patients embryos, discriminating between embryos with a normal set of chromosomes (euploid) and those with an abnormal set of chromosomes (aneuploid). In this study, we will apply a novel validated next generation sequencing technology called copy number variation sequencing (CNV-Seq) to comprehensively screen a trophectoderm biopsy sample from patient's embryos for chromosomal abnormalities that commonly arise in human embryos. The hypothesis is that PGS performed using CNV-Seq on embryos produced by patients with a poor prognosis for pregnancy (maternal age > 35), followed by transfer of chromosomally normal euploid embryos, will result in significantly higher implantation, pregnancy and live birth rates and lower miscarriage rates compared to patients having no PGS.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing in vitro fertilization (IVF)
* Normal uterine function by ultrasound and absence of hysteromyoma
* Regular menstrual cycle of 25-35 days
* Normal hormone levels (WHO standard) for LH, PRL, E2, PROG, TEST and TSH
* FSH 1-12 IU/L and follicle number > 5 on day 2-3 of menstrual cycle
* Minimum of 3 blastocysts on day 5 of embryo development
* Signed consent form

Exclusion Criteria:

* Known endometriosis
* Abnormal vaginal bleeding with no known cause
* Known genital organ system malformation, unsuitable to conceive
* Known currently active pelvic inflammation
* Abnormal liver, kidney lab results, with clinical implications.
* Known endocrine or metabolic disorders (pituitary gland, adrenal glands, pancreas, liver or kidney）
* Known ovarian, breast, uterine, adrenal glands, pituitary gland or hypothalamus tumor
* Known abnormal cervical cancer lesions, with clinical implications, within one year before PGS
* History of chemo- or radio-therapy
* Seropositive for HIV, Hep B, Hep C or TPPA/RPR (Syphilis)
* Known ovarian poor response in previous cycles, i.e. after administration of GnRH for > 20 days
* More than 2 implantation failures
* More than 2 miscarriages
* Known altered parental karyotype such as Robertsonian or reciprocal translocation
* Use of sperm or oocyte donors
* Severe male factor (surgical retrieval of sperm)
* Preimplantation genetic diagnosis cycles for single gene diseases or sex selection
* Participation in other IVF research studies
* Patient refusal or inability to follow the protocol for any good reason, including clinical visit or lab test

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-12 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy | Gestational week 20

SECONDARY OUTCOMES:
Genetic health of the fetus | Gestational week 18
  The patient will be offered a noninvasive prenatal test for fetal aneuploidies between 12-18 weeks gestation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Beijing, China

REFERENCES:
- [Background] Wang Y, Chen Y, Tian F, Zhang J, Song Z, Wu Y, Han X, Hu W, Ma D, Cram D, Cheng W. Maternal mosaicism is a significant contributor to discordant sex chromosomal aneuploidies associated with noninvasive prenatal testing. Clin Chem. 2014 Jan;60(1):251-9. doi: 10.1373/clinchem.2013.215145. Epub 2013 Nov 5. PMID 24193117
- [Background] Liang D, Peng Y, Lv W, Deng L, Zhang Y, Li H, Yang P, Zhang J, Song Z, Xu G, Cram DS, Wu L. Copy number variation sequencing for comprehensive diagnosis of chromosome disease syndromes. J Mol Diagn. 2014 Sep;16(5):519-526. doi: 10.1016/j.jmoldx.2014.05.002. Epub 2014 Jul 3. PMID 24998187
- [Background] Wang L, Wang X, Zhang J, Song Z, Wang S, Gao Y, Wang J, Luo Y, Niu Z, Yue X, Xu G, Cram DS, Yao Y. Detection of chromosomal aneuploidy in human preimplantation embryos by next-generation sequencing. Biol Reprod. 2014 May 8;90(5):95. doi: 10.1095/biolreprod.113.116459. Print 2014 May. PMID 24648399
- [Background] Wang L, Cram DS, Shen J, Wang X, Zhang J, Song Z, Xu G, Li N, Fan J, Wang S, Luo Y, Wang J, Yu L, Liu J, Yao Y. Validation of copy number variation sequencing for detecting chromosome imbalances in human preimplantation embryos. Biol Reprod. 2014 Aug;91(2):37. doi: 10.1095/biolreprod.114.120576. Epub 2014 Jun 25. PMID 24966395
- [Background] Wang H, Wang L, Ma M, Song Z, Zhang J, Xu G, Fan J, Li N, Cram DS, Yao Y. A PGD pregnancy achieved by embryo copy number variation sequencing with confirmation by non-invasive prenatal diagnosis. J Genet Genomics. 2014 Aug 20;41(8):453-6. doi: 10.1016/j.jgg.2014.06.007. Epub 2014 Jul 17. No abstract available. PMID 25160978
- [Derived] Cornelisse S, Zagers M, Kostova E, Fleischer K, van Wely M, Mastenbroek S. Preimplantation genetic testing for aneuploidies (abnormal number of chromosomes) in in vitro fertilisation. Cochrane Database Syst Rev. 2020 Sep 8;9(9):CD005291. doi: 10.1002/14651858.CD005291.pub3. PMID 32898291